CLINICAL TRIAL: NCT03570658
Title: A Randomized, Sponsor-Open, Investigator-Blinded, Subject-Blinded, Placebo-Controlled, Single-Ascending Dose (SAD) and Multiple-Ascending Dose (MAD) Study to Investigate the Safety, Tolerability, and Pharmacokinetics of RO7049389 in Healthy Chinese Subjects
Brief Title: A Double-Blind Single-Ascending Dose (SAD) and Multiple-Ascending Dose (MAD) Study to Investigate the Safety, Tolerability, and Pharmacokinetics of RO7049389 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: YP39406
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis B Virus
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-Ascending Dose (SAD) (Experimental): Participants will receive a single dose of RO7049389.
  Interventions: Drug: RO7049389
- Multiple-Ascending Dose (MAD) (Experimental): Participants will receive multiple doses of RO7049389.
  Interventions: Drug: RO7049389
- Placebo (Placebo Comparator): Participants will receive either a single dose (SAD cohorts) or multiple doses (MAD cohorts) of placebo matched to RO7049389.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7049389 — RO7049389 will be administered orally either as a single dose (SAD) or as multiple doses defined by the SAD portion of the study (MAD).
  Arms: Multiple-Ascending Dose (MAD); Single-Ascending Dose (SAD)
Drug: Placebo — Placebo will be administered orally at a dose and frequency matched to RO7049389.
  Arms: Placebo

SUMMARY:
This study will assess the safety and tolerability of RO7049389 compared to placebo in single- and multiple-ascending doses in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria

* Chinese healthy male and female subjects, 18 to 60 years of age, inclusive.
* A Body Mass Index (BMI) of between 19 to 27 kg/m2 inclusive, and a body weight of at least 45 kg.
* Women should be of non-childbearing potential. Female subjects must be either surgically sterile (by means of hysterectomy and/or bilateral oophorectomy) or post-menopausal for at least one year (defined as amenorrhea >/=12 consecutive months without another cause, and confirmed by follicle stimulating hormone level >35 mIU/mL).
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria

* Pregnant (positive pregnancy test) or lactating women, and male subjects with partners who are pregnant or lactating.
* History or symptoms of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis.
* Personal history of congenital long QT syndrome or family history of sudden death.
* History of Gilbert's syndrome.
* History of having received or currently receiving any systemic anti-neoplastic (including radiation) or immune-modulatory treatment (including systemic oral or inhaled corticosteroids) </=6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* Subjects who have had significant acute infection, e.g., influenza, local infection, acute gastrointestinal symptoms or any other clinically significant illness within two weeks of dose administration.
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable).
* Electrocardiogram (ECG) with QRS and/or T-wave judged to be unfavorable for a consistently accurate QT measurement (e.g., neuromuscular artifact that cannot be readily eliminated, arrhythmias, indistinct QTS onset, low amplitude T-wave, merged T- and U waves, prominent U-waves)
* Creatinine clearance (CrCl) </=70 mL/min (using the Cockcroft-Gault formula)
* Positive test at screening of any of the following: hepatitis A (HAV IgM Ab), hepatitis B (HBsAg), hepatitis C (HCV RNA or HCV Ab) or human immunodeficiency virus 1 and 2 (HIV Ab).
* Participation in an investigational drug or device study within 90 days prior to screening or more than 4 times per year.
* Donation or loss of blood over 500 mL within 3 months prior to screening.
* Any suspicion or history of drug and/or alcohol abuse within the last year.
* History (within 3 months of screening) of alcohol consumption exceeding two standard drinks per day on average (1 standard drink = 10 grams of alcohol). Alcohol consumption will be prohibited at least 48 hours before screening, 48 hours before and 48 hours after each dose, and 48 hours before each scheduled visit.
* Use of >5 cigarettes or equivalent nicotine-containing product per day.
* Taking any prescribed or over-the-counter medications (including vitamins or herbal remedies) within 2 weeks of first dosing or within 5 times the elimination half-life of the medication prior to first dosing (whichever is longer). Occasional acetaminophen/paracetamol is allowed.
* Subjects under judicial supervision, guardianship or curatorship.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China

REFERENCES:
- [Derived] Wu X, Feng S, Zhang J, Zhang W, Zhang Y, Zhu M, Triyatni M, Zhao N, Bo Q, Jin Y. Evaluation of the safety, tolerability, and pharmacokinetics of RO7049389 in healthy Chinese volunteers. Clin Transl Sci. 2022 Jan;15(1):195-203. doi: 10.1111/cts.13134. Epub 2021 Sep 25. PMID 34562067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male Chinese subjects aged 18-60 years.
Pre-assignment Details: Total n=31.
  SAD n=28 (Active treatment n=22 and placebo n=6). 21 participants continued on to the MAD phase of the study. 3 participants chose not to continue.
  MAD n=24. 3 participants were directly enrolled into the MAD phase of the study in addition to the 21 participants from the SAD phase.
Groups:
- Placebo: Participants in both the MAD and SAD cohorts received placebo matched to RO7049389.
- RO7049389 - 200 mg: Participants in the SAD cohort received a single 200 mg dose of RO7049389.
- RO7049389 - 400 mg/200 mg q12h: Participants in the SAD cohort received a single 400 mg dose of RO7049389. Participants in the MAD cohort that formerly received the 400 mg single dose received 200 mg of RO7049389 every 12 hours (q12h) for 14 days.
- RO7049389 - 600 mg/400 mg q12h: Participants in the SAD cohort only received a single 600 mg dose of RO7049389. Participants in the MAD cohort that formerly received the 600 mg single dose received 400 mg of RO7049389 q12h for 14 days.
Period: Single Ascending Dose (SAD)
Arm/Group | Placebo | RO7049389 - 200 mg | RO7049389 - 400 mg/200 mg q12h | RO7049389 - 600 mg/400 mg q12h
Started | 6 | 2 | 10 | 10
Completed | 6 | 2 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Multiple Ascending Dose (MAD)
Arm/Group | Placebo | RO7049389 - 200 mg | RO7049389 - 400 mg/200 mg q12h | RO7049389 - 600 mg/400 mg q12h
Started | 4 | 0 | 10 | 10
Completed | 4 | 0 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total n=31. SAD n=28. 21 participants continued and 3 new participants were directly enrolled in MAD (n=24). The 400/200 arm enrolled 2 new participants and the 600/400 arm enrolled 1. Baseline characteristics are split in to SAD and MAD to account for the 3 additional participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RO7049389 - 200 mg | RO7049389 - 400 mg/200 mg q12h | RO7049389 - 600 mg/400 mg q12h | Total
Number analyzed (Participants) | 6 | 2 | 12 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] — SAD participants Population: The SAD population included 28 participants assigned to either placebo or active treatment.
  Years
    number analyzed (Participants) | 6 | 2 | 10 | 10 | 28
    (all) | 29.2 (5.7) | 33.5 (6.4) | 30.2 (3.2) | 28.2 (6.0) | 29.5 (5.0)
Age, Continuous [Mean (Standard Deviation); unit: Years] — MAD participants Population: The MAD population included 24 participants assigned to either placebo or active treatment.
  Years
    number analyzed (Participants) | 4 | 0 | 10 | 10 | 24
    (all) | 28.8 (6.1) |  | 31.1 (3.3) | 29.0 (6.5) | 29.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants] — SAD participants Population: The SAD population included 28 participants assigned to either placebo or active treatment.
  Participants
    number analyzed (Participants) | 6 | 2 | 10 | 10 | 28
    Female | 0 | 0 | 0 | 0 | 0
    Male | 6 | 2 | 10 | 10 | 28
Sex: Female, Male [Count of Participants; unit: Participants] — MAD participants Population: The MAD population included 24 participants assigned to either placebo or active treatment.
  Participants
    number analyzed (Participants) | 4 | 0 | 10 | 10 | 24
    Female | 0 | 0 | 0 | 0 | 0
    Male | 4 |  | 10 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — SAD participants Population: The SAD population included 28 participants assigned to either placebo or active treatment.
  Participants
    number analyzed (Participants) | 6 | 2 | 10 | 10 | 28
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 6 | 2 | 10 | 10 | 28
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — MAD participants Population: The MAD population included 24 participants assigned to either placebo or active treatment.
  Participants
    number analyzed (Participants) | 4 | 0 | 10 | 10 | 24
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 4 | 0 | 10 | 10 | 24
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — SAD participants Population: The SAD population included 28 participants assigned to either placebo or active treatment.
  Participants
    number analyzed (Participants) | 6 | 2 | 10 | 10 | 28
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 6 | 2 | 10 | 10 | 28
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — MAD participants Population: The MAD population included 24 participants assigned to either placebo or active treatment.
  Participants
    number analyzed (Participants) | 4 | 0 | 10 | 10 | 24
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 4 | 0 | 10 | 10 | 24
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: From the date of first administered dose through 28 days after the last administered dose.
Population: All safety analyses were based on the safety analysis population, which included all subjects that received at least one dose of study medication (RO7049389 or placebo), with at least one safety assessment.
Measure: Number; unit: Percentage of Participants
Groups:
- SAD - Placebo; MAD - Placebo: Participants received placebo matched to RO7049389.
- SAD RO7049389 - 200 mg: Participants received a single 200 mg dose of RO7049389.
- SAD RO7049389 - 400 mg: Participants received a single 400 mg dose of RO7049389.
- SAD RO7049389 - 600 mg: Participants received a single 600 mg dose of RO7049389.
- MAD RO7049389 - 200 mg: Participants received 200 mg of RO7049389 every 12 hours for 14 days.
- MAD RO7049389 - 400 mg: Participants received 400 mg of RO7049389 every 12 hours for 14 days.
Arm/Group | SAD - Placebo | SAD RO7049389 - 200 mg | SAD RO7049389 - 400 mg | SAD RO7049389 - 600 mg | MAD - Placebo | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
Number analyzed (Participants) | 6 | 2 | 10 | 10 | 4 | 10 | 10
Percentage of Participants | 16.7 | 0 | 30.0 | 10.0 | 50.0 | 90.0 | 60.0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of RO7049389
Time Frame: At pre-defined intervals on Day 1 (SAD) and Day 14 (MAD)
Population: PK sampling was performed only once for single-dose (SAD) cohorts and did not include the placebo arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SAD RO7049389 - 200 mg | SAD RO7049389 - 400 mg | SAD RO7049389 - 600 mg | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
Number analyzed (Participants) | 2 | 10 | 10 | 10 | 10
ng/mL
  Day 1 | 3840 (41.3) | 5220 (84.8) | 4020 (116) | 3230 (40.6) | 9210 (51.1)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10
  Day 14 |  |  |  | 2730 (35.4) | 8030 (60.8)

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of RO7049389
Time Frame: At pre-defined intervals on Day 1 (SAD) and Day 14 (MAD)
Population: PK sampling was performed only once for single-dose (SAD) cohorts and did not include the placebo arms.
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | SAD RO7049389 - 200 mg | SAD RO7049389 - 400 mg | SAD RO7049389 - 600 mg | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
Number analyzed (Participants) | 2 | 10 | 10 | 10 | 10
Hours (h)
  Day 1 | 1.5 [1.5 to 1.5] | 1.5 [1 to 3] | 2 [1 to 4] | 1.5 [1.5 to 2] | 2 [1 to 3]
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10
  Day 14 |  |  |  | 2 [1.5 to 2.02] | 2 [1.5 to 3]

4. Secondary Outcome: Area Under the Plasma Concentration vs Time Curve to Last Measurable Concentration (AUClast) of RO7049389
Time Frame: At pre-defined intervals on Day 1 (SAD) and Day 14 (MAD)
Population: PK sampling was performed only once for single-dose (SAD) cohorts and did not include the placebo arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD RO7049389 - 200 mg | SAD RO7049389 - 400 mg | SAD RO7049389 - 600 mg | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
Number analyzed (Participants) | 2 | 10 | 10 | 10 | 10
h*ng/mL
  Day 1 | 5960 (60.9) | 12200 (85.1) | 10800 (121) | 5090 (38) | 19400 (72.6)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10
  Day 14 |  |  |  | 5460 (29.2) | 20900 (90.7)

5. Secondary Outcome: Area Under the Plasma Concentration vs Time Curve Extrapolated to Infinity (AUC0-inf)
Time Frame: At pre-defined intervals on Day 1 (SAD) and Day 14 (MAD)
Population: PK sampling was performed only once for single-dose (SAD) cohorts and did not include the placebo arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD RO7049389 - 200 mg | SAD RO7049389 - 400 mg | SAD RO7049389 - 600 mg | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
Number analyzed (Participants) | 2 | 10 | 10 | 10 | 10
h*ng/mL
  Day 1: number analyzed (Participants) | 1 | 10 | 9 | 10 | 10
  Day 1 | 9460 (NA) — NA = there was only one participant sample. | 12300 (84.6) | 11100 (120) | 5180 (37.7) | 19500 (72.7)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10
  Day 14 |  |  |  | 5470 (29.1) | 20900 (90.6)

6. Secondary Outcome: Apparent Half-Life (T1/2) of RO7049389
Time Frame: At pre-defined intervals on Day 1 (SAD) and Day 14 (MAD)
Population: PK sampling was performed only once for single-dose (SAD) cohorts and did not include the placebo arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | SAD RO7049389 - 200 mg | SAD RO7049389 - 400 mg | SAD RO7049389 - 600 mg | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
Number analyzed (Participants) | 2 | 10 | 10 | 10 | 10
Hours (h)
  Day 1: number analyzed (Participants) | 1 | 10 | 9 | 10 | 10
  Day 1 | 3.66 (0) | 7.98 (97.8) | 10.4 (108) | 2.29 (39.4) | 1.62 (33.1)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10
  Day 14 |  |  |  | 5.06 (31.6) | 6.74 (36.4)

7. Secondary Outcome: Clearance (CL/F) of RO7049389
Time Frame: At pre-defined intervals on Day 1 (SAD)
Population: This parameter was not collected for the MAD cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | SAD RO7049389 - 200 mg | SAD RO7049389 - 400 mg | SAD RO7049389 - 600 mg
Number analyzed (Participants) | 2 | 10 | 10
L/h | 21.1 (0) | 32.6 (58.2) | 53.9 (61.8)

8. Secondary Outcome: Trough Plasma Concentration (Ctrough) of RO7049389
Time Frame: At pre-defined intervals on Day 14 (MAD)
Population: This outcome measure applied to arms receiving RO7049389 during the MAD phase.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
Number analyzed (Participants) | 10 | 10
ng/mL | 31.1 (29.8) | 66.1 (133)

9. Secondary Outcome: Accumulation Index of RO7049389
Time Frame: At pre-defined intervals on Day 14 (MAD)
Population: This parameter was not collected for SAD cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
Number analyzed (Participants) | 10 | 10
Ratio
  MAD Cohorts - Day 14 Cmax | 0.846 (76.9) | 0.872 (41.7)
  MAD Cohorts - Day 14 AUC | 1.03 (47) | 1.05 (37.6)

10. Secondary Outcome: Area Under the Concentration vs Time Curve for a Dosing Interval (AUCtau)
Time Frame: At pre-defined intervals on Day 14 (MAD)
Population: This parameter was not collected for SAD cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- RO7049389 - 400 mg: Participants in the SAD cohort received a single 400 mg dose of RO7049389, followed by a 1-week washout period. Participants in the MAD cohort that formerly received the 600 mg single dose received 400 mg of RO7049389 every 12 hours for 14 days.
Arm/Group | MAD RO7049389 - 200 mg | RO7049389 - 400 mg
Number analyzed (Participants) | 10 | 10
h*ng/mL
  MAD Cohorts - Day 1 | 5090 (38) | 19400 (72.6)
  MAD Cohorts - Day 14 | 5230 (29.7) | 20400 (90.7)

ADVERSE EVENTS:
Time Frame: From the date of first administered dose through 28 days after the last administered dose.
Arm/Group | SAD - Placebo | SAD RO7049389 - 200 mg | SAD RO7049389 - 400 mg | SAD RO7049389 - 600 mg | MAD - Placebo | MAD RO7049389 - 200 mg | MAD RO7049389 - 400 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/10 | 0/10 | 0/4 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/10 | 0/10 | 0/4 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 0/2 | 3/10 | 1/10 | 2/4 | 9/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAD - Placebo (N=6) | SAD RO7049389 - 200 mg (N=2) | SAD RO7049389 - 400 mg (N=10) | SAD RO7049389 - 600 mg (N=10) | MAD - Placebo (N=4) | MAD RO7049389 - 200 mg (N=10) | MAD RO7049389 - 400 mg (N=10)
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Eosinophil percentage increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary casts present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 8 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT03570658/Prot_SAP_000.pdf